CLINICAL TRIAL: NCT01188187
Title: A Randomized Phase 3 Study Comparing Standard First-Line Docetaxel/Prednisone to Docetaxel/Prednisone in Combination With Custirsen (OGX-011) in Men With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Comparison of Docetaxel/Prednisone to Docetaxel/Prednisone in Combination With OGX-011 in Men With Prostate Cancer
Acronym: SYNERGY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGX-011-11 TRANSFERRED
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: custirsen sodium; prostate cancer; overall survival; Metastatic Castrate Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — OGX-011; Docetaxel; Prednisone; Dexamethasone

ARMS (2):
- Custirsen, Docetaxel, Prednisone (Experimental): Three doses of 640 mg custirsen administered intravenously (IV) as a loading dose between Days -9 to -1. Custirsen, 640 mg, given IV weekly on Days 1, 8, and 15 of each 21-day cycle. Docetaxel (75 mg/M^2 via intravenous injection) on Day 1 of every 21 days plus prednisone (5 mg tablets taken by mouth) twice each day and dexamethasone (8 mg by mouth twice a day for 3 days beginning one day before docetaxel administration).
  Treatment continues for 10 cycles or until unacceptable toxicity or disease progression.
  Interventions: Drug: Custirsen; Drug: Docetaxel; Drug: Prednisone; Drug: Dexamethasone
- Docetaxel, Prednisone (Active Comparator): Docetaxel (75 mg/M^2 via intravenous injection) on Day 1 of every 21 days plus prednisone (5 mg tablets taken by mouth) twice each day and dexamethasone (8 mg by mouth twice a day for 3 days beginning one day before docetaxel administration).
  Treatment continues for 10 cycles or until unacceptable toxicity or disease progression.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Dexamethasone

INTERVENTIONS:
Drug: Custirsen
  Other Names: OGX-011
  Arms: Custirsen, Docetaxel, Prednisone
Drug: Docetaxel
Drug: Prednisone
Drug: Dexamethasone — Dexamethasone 8 mg by mouth twice a day for 3 days beginning one day before docetaxel administration to reduce the incidence and severity of hypersensitivity reactions and fluid retention.

SUMMARY:
This Phase 3 study has been designed to confirm that adding custirsen to standard first-line docetaxel/prednisone treatment can slow tumor progression and enhance survival outcomes compared to standard first-line docetaxel/prednisone treatment alone. This will be a randomized, open-label, multicenter, international trial. Treatment will consist of docetaxel/prednisone/custirsen vs. docetaxel/prednisone. A total of at least 1000 patients will be randomized. Patients will be randomly assigned with equal probability to the two arms.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years on the date of consent.
* Histological or cytological diagnosis of adenocarcinoma of the prostate.
* Metastatic disease on chest, abdominal, or pelvic CT and/or bone scan.
* Systemic chemotherapy indicated due to progression while on or after androgen ablative therapy defined as:

  1. Progressive measurable disease: at least a 20% increase in the sum of the longest diameters of measurable lesions over the smallest sum observed -or- the appearance of one or more new lesions as assessed by CT scan during hormone ablation treatment. Measurable lesions are nodal or visceral soft-tissue lesions with nodal lesions ≥ 20 mm in diameter or visceral/soft-tissue lesions ≥ 10 mm in diameter (see Section 6.3.1.1 ).

     OR
  2. Bone Scan Progression: appearance of 2 or more new lesions on bone scan during hormone ablation treatment.

     OR
  3. Increasing serum prostate-specific antigen (PSA) level: Two consecutive increases in PSA levels documented over a previous reference value obtained at least one week apart are required. If the third PSA value is less than the second, an additional fourth test to confirm a rising PSA is acceptable. A minimum starting value of 5.0 ng/mL is required for study randomization.
* Baseline laboratory values as stated below:

  1. Creatinine ≤ 1.5 x upper limit of normal (ULN).
  2. Bilirubin ≤ 1.1 x ULN (unless elevated secondary to conditions such as Gilbert's disease).
  3. Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) ≤ 1.5 x ULN.
  4. Castrate serum testosterone level (< 50 ng/dL-or-< 1.7 nmol/L).
* Must be willing to continue primary androgen suppression with gonadotropin-releasing hormone (GnRH) analogues (either agonists or antagonists) throughout the study, unless treated with bilateral orchiectomy.
* Adequate bone marrow function defined at screening as absolute neutrophil count (ANC) ≥ 1.5 x 10^9 cells /L and platelet count ≥ 100 x 10^9 /L.
* Karnofsky score ≥ 70% (see Appendix 17.2).
* At least 28 days has passed since completing radiotherapy (exception for radiotherapy: at least 7 days since completing a single fraction of ≤ 800 centigray (cGy) to a restricted field or limited-field radiotherapy to non-marrow bearing area such as an extremity or orbit) at the time of randomization.
* At least 4 weeks have passed since receiving any investigational agent at the time of randomization.
* Has recovered from any other therapy-related toxicity to ≤ grade 2, (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy).
* Patient must be willing to not add, delete or change their current bisphosphonate or denosumab usage throughout study treatment to assure that adverse event reporting is not confounded by changing their bisphosphonate or denosumab usage (unless withdrawn or changed as a result of bisphosphonate or denosumab associated toxicity).
* Patients receiving more than 10 mg of prednisone per day (or steroid equivalent) at screening must be willing to have the dose reduced to 10 mg of prednisone per day for at least 7 days prior to randomization and maintained throughout study treatment.
* Written informed consent must be obtained prior to any protocol-specific procedures being performed.

Exclusion Criteria

* Received any other cytotoxic chemotherapy as treatment for prostate cancer.
* Received any cycling, intermittent or continuous hormonal treatment 28 days prior to randomization with the exception of the continuous GnRH analogues required in Inclusion Criteria #6.
* Participated in a prior clinical study evaluating custirsen.
* History of or current documented brain metastasis or carcinomatous meningitis, treated or untreated. (Brain imaging for asymptomatic patients is not required.)
* Current symptomatic cord compression requiring surgery or radiation therapy. (Once successfully treated and there has been no progression, patients are eligible for the study.) -Active second malignancy (except non-melanomatous skin or superficial bladder cancer) defined as requiring anticancer therapy or at high risk of recurrence during the study.
* Active second malignancy (except non melanomatous skin or superficial bladder cancer) defined as requiring cancer therapy or at high risk of reoccurrence during the study
* Uncontrolled medical conditions such as heart failure, myocardial infarction, uncontrolled hypertension, stroke or treatment of a major active infection within 3 months of randomization, as well as any significant concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy.
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device. Concomitant participation in observational studies is acceptable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier Estimates for Time to Death (Overall Survival) | Randomization (approximately Day -12) to longest survival follow-up (Day 971).
  Time from the date of randomization to death from any cause. After stopping treatment, patients were followed every 4 weeks until disease progression and then followed every 12 weeks until death.

SECONDARY OUTCOMES:
Percentage of Participants Who Were Alive Without Event At Day 140 | Day 125-155
  Patients who were alive without event (AWE) are patients who had their Milestone Day 140 Disease Status performed per protocol (Day 125 - Day 155 window), were not determined to have disease progression by the investigator on that window and confirmed as not having progressive disease (NONPD) by the Central Imagine Lab independent review.
Percentage of Participants with Adverse Events | Docetaxel/prednisone/custirsen arm: Days -9 up to Day 743. Docetaxel/prednisone arm: Day 1 up to Day 400.
  An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the administration, at any dose, of a medicinal or therapeutic product whether or not considered related to that product. Severity was rated by the investigator on a scale of 1 (mild) to 5 (death). A severity of 3 = Severe or medically significant but not immediately life-threatening. A severity of 4 = Life-threatening. Serious AEs include death (death due to progressive disease were not reported as an SAE), a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Celestia Higano, MD, Study Chair — Seattle Cancer Care Alliance, US; Kim Chi, MD, Study Chair — Vancouver Prostate Centre, BC Cancer Agency, Canada; Johann de Bono, Professor, Study Chair — Institute of Cancer Research, UK
Locations (140):
- United States (25):
  - Teva Investigational Site 100, Birmingham, Alabama
  - Teva Investigational Site 086, Los Angeles, California
  - Teva Investigational Site 263, Los Angeles, California
  - Teva Investigational Site 093, Marina del Rey, California
  - Teva Investigational Site 097, San Diego, California
  - Teva Investigational Site 090, Fort Collins, Colorado
  - Teva Investigational Site 106, Fort Myers, Florida
  - Teva Investigational Site 094, Port Saint Lucie, Florida
  - Teva Investigational Site 096, Atlanta, Georgia
  - Teva Investigational Site 103, Baton Rough, Louisiana
  - Teva Investigational Site 098, Ann Arbor, Michigan
  - Teva Investigational Site 112, Detroit, Michigan
  - Teva Investigational Site 032, Rochester, Minnesota
  - Teva Investigational Site 204, Las Vegas, Nevada
  - Teva Investigational Site 107, Cincinnati, Ohio
  - Teva Investigational Site 266, Greensboro, South Carolina
  - Teva Investigational Site 102, Myrtle Beach, South Carolina
  - Teva Investigational Site 084, Memphis, Tennessee
  - Teva Investigational Site 101, Nashville, Tennessee
  - Teva Investigational Site 116, San Antonio, Texas
  - Teva Investigational Site 059, Tyler, Texas
  - Teva Investigational Site 063, Tyler, Texas
  - Teva Investigational Site 047, Newport, Virginia
  - Teva Investigational Site 104, Norfolk, Virginia
  - Teva Investigational Site 029, Seattle, Washington
- Belgium (4):
  - Teva Investigational Site 862, Bonheiden
  - Teva Investigational Site 860, Brussels
  - Teva Investigational Site 864, Edegem
  - Teva Investigational Site 863, Ghent
- Canada (16):
  - Teva Investigational Site 002, Calgary, Alberta
  - Teva Investigational Site 023, Edmonton, Alberta
  - Teva Investigational Site 118, Abbotsford, British Columbia
  - Teva Investigational Site 007, Surrey, British Columbia
  - Teva Investigational Site 001, Vancouver, British Columbia
  - Teva Investigational Site 085, Victoria, British Columbia
  - Teva Investigational Site 024, Winnipeg, Manitoba
  - Teva Investigational Site 028, Halifax, Nova Scotia
  - Teva Investigational Site 025, Hamilton, Ontario
  - Teva Investigational Site 108, Kingston, Ontario
  - Teva Investigational Site 091, Oshawa, Ontario
  - Teva Investigational Site 003, Ottawa, Ontario
  - Teva Investigational Site 004, Toronto, Ontario
  - Teva Investigational Site 087, Toronto, Ontario
  - Teva Investigational Site 026, Montreal, Quebec
  - Teva Investigational Site 027, Montreal, Quebec
- France (14):
  - Teva Investigational Site 551, Angers
  - Teva Investigational Site 552, Avignon
  - Teva Investigational Site 553, Grenoble
  - Teva Investigational Site 555, La Roche-sur-Yon
  - Teva Investigational Site 557, Marseille
  - Teva Investigational Site 558, Nice
  - Teva Investigational Site 559, Paris
  - Teva Investigational Site 560, Paris
  - Teva Investigational Site 566, Saint-Brieuc
  - Teva Investigational Site 561, Saint-Herblain
  - Teva Investigational Site 562, Saint-Priest-en-Jarez
  - Teva Investigational Site 563, Toulouse
  - Teva Investigational Site 564, Vandœuvre-lès-Nancy
  - Teva Investigational Site 550, Villejuif
- Germany (19):
  - Teva Investigational Site 607, Aachen
  - Teva Investigational Site 609, Berlin
  - Teva Investigational Site 613, Berlin
  - Teva Investigational Site 604, Darmstadt
  - Teva Investigational Site 612, Dresden
  - Teva Investigational Site 618, Greifswald
  - Teva Investigational Site 600, Hanover
  - Teva Investigational Site 606, Heidelberg
  - Teva Investigational Site 615, Heinsberg
  - Teva Investigational Site 611, Homburg/Saar
  - Teva Investigational Site 617, Kempen
  - Teva Investigational Site 608, Marburg
  - Teva Investigational Site 616, Meiningen
  - Teva Investigational Site 614, München
  - Teva Investigational Site 601, Münster
  - Teva Investigational Site 602, Nürtingen
  - Teva Investigational Site 603, Stuttgart
  - Teva Investigational Site 610, Tübingen
  - Teva Investigational Site 605, Wuppertal
- Hungary (9):
  - Teva Investigational Site 691, Budapest
  - Teva Investigational Site 694, Budapest
  - Teva Investigational Site 692, Debrecen
  - Teva Investigational Site 697, Debrecen
  - Teva Investigational Site 696, Győr
  - Teva Investigational Site 698, Miskolc
  - Teva Investigational Site 699, Nyíregyháza
  - Teva Investigational Site 693, Szeged
  - Teva Investigational Site 695, Veszprém
- Israel (6):
  - Teva Investigational Site 506, Jerusalem, IL
  - Teva Investigational Site 507, Haifa
  - Teva Investigational Site 505, Petah Tikva
  - Teva Investigational Site 502, Ramat Gan
  - Teva Investigational Site 503, Tel Aviv
  - Teva Investigational Site 501, Zrifin
- Italy (14):
  - Teva Investigational Site 753, Arezzo
  - Teva Investigational Site 758, Catanzaro
  - Teva Investigational Site 760, Cesena (FC)
  - Teva Investigational Site 752, Genova
  - Teva Investigational Site 755, Lugo (Ravenna)
  - Teva Investigational Site 759, Meldola (FC)
  - Teva Investigational Site 763, Milan
  - Teva Investigational Site 754, Napoli
  - Teva Investigational Site 756, Napoli
  - Teva Investigational Site 761, Rimini
  - Teva Investigational Site 750, Roma
  - Teva Investigational Site 762, Roma
  - Teva Investigational Site 764, Rozzano (MI)
  - Teva Investigational Site 765, Verona
- Netherlands (3):
  - Teva Investigational Site 851, Amsterdam
  - Teva Investigational Site 852, Rotterdam
  - Teva Investigational Site 853, Sittard-Geleen
- South Korea (7):
  - Teva Investigational Site 404, Cheongju,Chungbuk
  - Teva Investigational Site 401, Goyang-si Gyeonggi-do
  - Teva Investigational Site 400, Seoul
  - Teva Investigational Site 402, Seoul
  - Teva Investigational Site 403, Seoul
  - Teva Investigational Site 406, Seoul
  - Teva Investigational Site 405, Yangsan
- Spain (16):
  - Teva Investigational Site 803, Barcelona
  - Teva Investigational Site 808, Barcelona
  - Teva Investigational Site 809, Barcelona
  - Teva Investigational Site 816, Dos Hermanas
  - Teva Investigational Site 814, El Palmar
  - Teva Investigational Site 807, Guadalajara
  - Teva Investigational Site 800, Madrid
  - Teva Investigational Site 801, Madrid
  - Teva Investigational Site 806, Madrid
  - Teva Investigational Site 813, Madrid
  - Teva Investigational Site 815, Manresa
  - Teva Investigational Site 810, Murcia
  - Teva Investigational Site 811, Palma de Mallorca
  - Teva Investigational Site 805, Pamplona
  - Teva Investigational Site 804, Sabadell - Barcelona
  - Teva Investigational Site 802, Valencia
- United Kingdom (7):
  - Teva Investigational Site 704, Brighton
  - Teva Investigational Site 701, Cambridge
  - Teva Investigational Site 709, Coventry
  - Teva Investigational Site 705, Guildford, Surrey
  - Teva Investigational Site 703, Manchester
  - Teva Investigational Site 710, Metropolitan Borough of Wirral
  - Teva Investigational Site 700, Surrey

REFERENCES:
- [Derived] Chi KN, Higano CS, Blumenstein B, Ferrero JM, Reeves J, Feyerabend S, Gravis G, Merseburger AS, Stenzl A, Bergman AM, Mukherjee SD, Zalewski P, Saad F, Jacobs C, Gleave M, de Bono JS. Custirsen in combination with docetaxel and prednisone for patients with metastatic castration-resistant prostate cancer (SYNERGY trial): a phase 3, multicentre, open-label, randomised trial. Lancet Oncol. 2017 Apr;18(4):473-485. doi: 10.1016/S1470-2045(17)30168-7. Epub 2017 Mar 8. PMID 28283282
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180